CLINICAL TRIAL: NCT04234958
Title: Études Des Effets d'un Protocol de thérapie Manuelle ostéopathique Sur la variabilité de la fréquence Cardiaque
Brief Title: Short- and Long-term HRV Measurements After Osteopathic Myofascial Thoracic Manipulations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec a Montréal (Other)
Collaborators: Collège d'Études Ostéopathiques de Montreal (Unknown)
Responsible Party: Principal Investigator, Alain Steve Comtois, Professor, Université du Québec a Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UQAMCEO_01
Record Dates: First submitted 2020-01-15; First posted 2020-01-21 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Heart Rate Variability
Keywords: heart rate variability; autonomous nervous system; osteopathy; osteopathy manipulative treatment; visceral; pericardium
MeSH Terms: interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental (Experimental): Participants received osteopathic treatment
  Interventions: Other: Osteopathic manipulative treatment
- Sham (Sham Comparator): Participants received sham therapy
  Interventions: Other: Sham therapy
- Control (No Intervention): Participants received no intervention

INTERVENTIONS:
Other: Osteopathic manipulative treatment — Specific protocol including 4 osteopathic techniques targeting the pericardium
  Arms: Experimental
Other: Sham therapy — Sham therapy mimicking the osteopathic techniques applied to experimental group
  Arms: Sham

SUMMARY:
The adaptation of the heart to react to any stimulus is called heart rate variability (HRV). Moreover, HRV is now used as a health index. In fact, among the pathologies affecting HRV the most, there are the cardiovascular diseases and depressive disorders that take a predominant part in the investigator's actual societies, According to a recent literature overview, many factors influence HRV and they need to be determined in order to plan efficient research protocols. Moreover, the control of these factors can improve the HRV and therefore help the heart to have maximum capacity to fulfill its physiological functions. Valorizing a good HRV seems, according to the effects reported by several studies, to be a good opportunity to take into consideration and to apply.

Visceral osteopathy, even if it goes back to the founder of Osteopathy himself, Andrew Taylor Still, is at its debuts in terms of acknowledgement from a scientific point of view. The evidence of efficacy of osteopathy is not to be done anymore. However, it is now necessary to define the action mechanisms of the osteopathic techniques, particularly by using physiological variables, and starting from a biomechanical angle. In fact, Jean-Pierre Barral and others has developed visceral manipulation techniques based on the viscera anatomy.

The originality of this research can be found in the technical protocol, not used yet, the use of witness group, the measurements over four weeks to evaluate the effect of this protocol with time on chosen dependant variables, its reproducibility but also its inter-therapist variance. This objective if this study is to reinforce the proof level of the osteopathic approach on the cardiac physiology. HRV is a solid tool recognized for research, the variable is well isolated and the control group ensures an isolation of some confounding variables.

ELIGIBILITY:
Inclusion Criteria:

* man or woman
* between 25 and 35 years old
* healthy
* non smoking

Exclusion Criteria:

* diagnosed with anxiety or psychological disorder
* smoker, drug consumption
* diagnosed with renal disorder, cardiac disorder, functional somatic disorders, diabetes, chronic alcoholism, cancer or immunosuppressive disorders, stroke, aortic aneurysm,
* pregnant
* high level athletes
* thoracic trauma or surgeries
* does not fit Hexoskin vest for HRV measurements
* does not complete all sessions
* cannot stay lying down for 1 hour
* below 25 or above 35 years old
* student in manual therapy

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-01-17 (Actual); Study Completion 2018-01-17 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | 45 minutes
  Real-time measurements of HRV before, during and after each intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Collège d'Études Ostéopathiques, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No